CLINICAL TRIAL: NCT06786637
Title: A Combined Investigation of the Protective Impact of the NOF/Q Antagonist LY-2940094 on Stress-induced Depression- and Anxiety-related Phenotypes in Humans
Brief Title: Investigating the Protective Impact of LY-2940094 on Stress-induced Depression- and Anxiety-related Phenotypes in Humans
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI transferred to a different research institution and local institution would not allow to continue the study. Transfer of the study to a different study site not possible because of unique requirements of resources (e.g., nociceptin anatagonist)
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Manuel Kuhn, Instructor, Department of Psychiatry, Harvard Medical School, McLean Hospital, McLean Hospital, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023A062574; 5P50MH119467-05 (NIH)
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder; Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders | interventions — LY2940094

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants receiving the nociceptin receptor antagonist (Experimental): After a diagnostic interview during the first visit, participants will receive the nociceptin receptor antagonist (LY-2940094) at the beginning of the second visit. Participants will then complete two computerized tasks (the Probabilistic Rewards Task (PRT) and a context fear conditioning paradigm). Tasks will begin 2 hours after the nociceptin receptor antagonist is administered.
  Interventions: Drug: Nociceptin Receptor Antagonist (LY-2940094); Device: DS8R Biphasic Constant Current Stimulator
- Participants receiving the placebo (Placebo Comparator): After a diagnostic interview during the first visit, participants will receive the placebo at the beginning of the second visit. Participants will then complete two computerized tasks (the Probabilistic Rewards Task (PRT) and a context fear conditioning paradigm). Tasks will begin 2 hours after the placebo is administered.
  Interventions: Device: DS8R Biphasic Constant Current Stimulator

INTERVENTIONS:
Drug: Nociceptin Receptor Antagonist (LY-2940094) — Participants in the experimental arms will receive 40 mg of the nociceptin receptor antagonist LY-2940094. Peak concentrations are achieved 2-4 hours post-administration.
  Other Names: Nociceptin Receptor Antagonist (BTRX-246040); Nociceptin Receptor Antagonist (C220614004-FP)
  Arms: Participants receiving the nociceptin receptor antagonist
Device: DS8R Biphasic Constant Current Stimulator — As part of the fear conditioning task, electrotactile stimulation will be used. The aversive stimulus is delivered in the form of a mild half-second stimulation to the ankle, calibrated to a subjective threshold that is uncomfortable but not painful. This stimulation is delivered by Digitimer DS8R Constant Current Stimulator (Digitimer North America, LLC. Ft. Lauderdale, FL). This model has been safely implemented in studies within McLean Hospital and Massachusetts General Hospital.

SUMMARY:
This project will integrate pharmacological and psychophysiological methodology to mechanistically investigate, in humans, the role of N/OFQ in laboratory phenotypes of both disorders. Specifically, a N/OFQ receptor (NOPR) antagonist will be used to test the hypothesis that NOPR blockage will have antidepressant-like effects (potentiate reward processing); in addition, this study will also evaluate a key anxiety phenotype (fear learning). Finally, the impact of recent life stress on these processes will be assessed. Results will demonstrate the specificity of NOPR blockage on depressive phenotypes or suggest a common pathway for emotional disorders and will confirm a modulatory role of life stress.

ELIGIBILITY:
Inclusion Criteria:

* Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse), as assessed by subject history and a structured clinical interview (diagnosed using the SCID-5)
* Written informed consent
* Absence of any medications for at least 3 weeks

Exclusion Criteria:

* Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician
* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder
* History or current diagnosis of any of the following DSM-IV psychiatric illnesses: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, obsessive-compulsive disorder, patients with mood congruent or mood incongruent psychotic features, substance dependence, substance abuse within the last 12 months (with the exception of cocaine or stimulant abuse; which will lead to exclusion)
* History of cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine)
* History of use of dopaminergic drugs (including methylphenidate)
* History or current diagnosis of dementia
* Patients with mood congruent or mood incongruent psychotic features
* Current use of other psychotropic drugs
* Clinical or laboratory evidence of hypothyroidism
* Patients with a lifetime history of electroconvulsive therapy
* Abnormal ECG and lab results
* History of seizure disorder or currently on anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (SCID-5) | Baseline
  The Structured Clinical Interview for DSM-5 (SCID-5) is a clinician-administered diagnostic tool used to assess and diagnose mental disorders based on DSM-5 criteria. The SCID-5 categorically identifies the presence or absence of specific diagnoses and does not provide numerical minimum/maximum values.
Childhood Trauma Questionnaire (CTQ) | Baseline
  The Childhood Trauma Questionnaire (CTQ) is a self-report tool assessing childhood emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Scores on each subscale range from 5 to 25, with a total score ranging from 25 to 125; higher scores indicate greater severity of childhood trauma.
List of Threatening Experiences Questionnaire (LTE) | Baseline
  The List of Threatening Experiences Questionnaire (LTE) is a self-report measure assessing the occurrence of stressful life events, such as bereavement, illness, or job loss, over a specified period. Scores range from 0 to 12, representing the number of endorsed events, with higher scores indicating a greater number of stressful experiences.
Combined Cue-Context Fear Conditioning Task: Subjective Fear Ratings | Baseline
  The combined cue-context fear conditioning task is a paradigm to assess fear learning and extinction in response to discrete cues as well as different contexts. Subjective ratings of fear are collected via visual analog scales throughout the task. Higher ratings mean higher expression of fear towards cues and contexts (min-max: 0-100).
Probabilistic Reward Task (PRT) | Baseline
  The Probabilistic Reward Task (PRT) is a behavioral measure assessing reward sensitivity and reinforcement learning. It evaluates participants' ability to modulate behavior based on probabilistic feedback associated with correct responses. The primary outcome is the response bias score, which ranges from negative values to positive values. Higher scores indicate a stronger bias toward the more frequently rewarded response, reflecting greater reward sensitivity and reinforcement learning. Lower or negative scores suggest impaired reward responsiveness, which is often associated with anhedonia or mood disorders.
Perceived Stress Scale | Baseline
  The Perceived Stress Scale (PSS) is a self-report measure assessing the degree to which situations in life are perceived as stressful over the past month. Scores range from 0 to 40, with higher scores indicating greater perceived stress.
Combined Cue-Context Fear Conditioning Task: Skin Conductance Responce (SCR) | Baseline
  The combined cue-context fear conditioning task is a paradigm to assess fear learning and extinction in response to discrete cues as well as different contexts. Skin conductance response (SCR) is a psychophysiological measure assessing objective levels of arousal. Skin conductance is measured in microsiemens (µS) and will be processed to quantify amplitude changes in response to task stimuli. Higher amplitudes indicate higher arousal levels in response to task stimuli (min: 0, max: none).
Combined Cue-Context Fear Conditioning Task: Fear-Potentiated Startle (FPS) | Baseline
  The combined cue-context fear conditioning task is a paradigm to assess fear learning and extinction in response to discrete cues as well as different contexts. Fear-potentiated startle (FPS) is a psychophysiological measure assessing objective levels of fear responses. FPS is a difference score between threat stimuli and neutral stimuli, both measured in microvolts (µV) and processed to quantify amplitude changes, in response to task stimuli. Higher FPS scores indicate higher fear levels towards the threat stimuli (min: none, max: none).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Kuhn, Ph.D., Principal Investigator — Mclean Hospital

IPD SHARING:
Plan to Share IPD: Yes
Through NIMH Data Archive and ClinicalTrials.gov, we will share the primary and secondary outcomes.